

# 6009-CONT Clinical Protocol

# Consumer Evaluation of Intermittent Catheter Product Modifications

Protocol Release Date: April 13, 2021 NCT04619992

#### **STUDY SPONSOR**

Hollister Incorporated 2000 Hollister Drive | Libertyville, IL 60048 | USA

Company Confidential: No portion of this work may be reproduced in whole or in part without the express written permission of Hollister Incorporated. This document contains confidential information for use only by individuals participating in the study or evaluation. This document should be maintained in a secure location and should not be copied or made available for review by any unauthorized person or firm. Copyright 2020 Hollister Incorporated.

Caution: Investigational device, limited by Federal (US) law to investigational use.

## **TABLE OF CONTENTS**

| 1.0 | ABRE | VIATIONS AND TERMS | 4 |
|---|---|---|---|
| 2.0 | ETHIC | CS | 5 |
| | 2.1 | IRB Review | 5 |
| | 2.2 | Name and Address of IRB | 5 |
| | 2.3 | Adherence to Ethical Principles | 5 |
| 3.0 | INVES | STIGATORS AND STUDY ADMINISTRATIVE STRUCTURE | 5 |
| | 3.1 | Investigator Responsibilities | 5 |
| | 3.2 | Sponsor Responsibilities | 5 |
| 4.0 | BACK | GROUND/RATIONALE | 6 |
| 5.0 | STUD | Y OBJECTIVES | 6 |
| | 5.1 | Primary Objective | 6 |
| | 5.2 | Secondary Objective | 6 |
| 6.0 | STUD | Y PRODUCTS | 6 |
| | 6.1 | Investigational Devices | 6 |
| | 6.2 | Identity of Product, Packaging and Storage, Procedures for Release | 7 |
| | 6.3 | Responsibility for Product Control, Return, and Disposal | 8 |
| 7.0 | STUD | Y DESIGN | 9 |
| 8.0 | STUD | Y SUBJECTS | 10 |
| | 8.1 | Inclusion Criteria for Group 1 | 10 |
| | 8.2 | Inclusion Criteria for Group 2 | 10 |
| | 8.3 | Exclusion Criteria for Group 1 | 11 |
| | 8.4 | Exclusion Criteria for Group 2 | 11 |
| | 8.5 | Subject Treatment and Care | 11 |
| | 8.6 | Subject Compensation | 11 |
| 9.0 | STUD | Y PROCEDURES | 12 |
| | 9.1 | Subject Identification and Recruitment | 12 |
| | 9.2 | Informed Consent | 12 |
| | 9.3 | Enrollment | 12 |
| | 9.4 | Method of Assigning Subjects to Study Groups | 13 |
| | 9.5 | Blinding | 13 |
| | 9.6 | Prior and Concomitant Therapy | 13 |
| | 9.7 | Study Visits and Evaluation Methods | 13 |
| | 9.8 | Subject Instructions | 16 |
| | 9.9 | Compliance | 16 |

| | 9.10 | Subject Withdrawal | 16 |
|---|---|---|---|
| 10.0 | ADVERSE EVENTS | | 17 |
| | 10.1 | Handling Adverse Events | 17 |
| | 10.2 | Reporting Adverse Events | 18 |
| | 10.3 | Study Stopping Rules | 18 |
| 11.0 | DATA | MANAGEMENT | 18 |
| 12.0 | STATIS | STICAL METHODS | 19 |
| | 12.1 | Analysis Principles | 19 |
| | 12.2 | Incomplete Follow-up and Missing Data | 19 |
| | 12.3 | Multi-Center and Multiple Comparison/Multiplicity Adjustments | 19 |
| | 12.4 | Sample Size and Power | 19 |
| 13.0 | STATIS | STICAL ANALYSES | 19 |
| | 13.1 | Primary and Secondary Objective | 19 |
| | 13.2 | Interim Analyses | 19 |
| 14.0 | STUD | OOCUMENTATION AND RECORD KEEPING | 20 |
| 15.0 | FINAL | REPORT | 20 |
| 16.0 | MONI | TORING | 20 |
| 17.0 | AMEN | DMENT PROCEDURES | 20 |
| 18.0 | PROT | DCOL ATTACHMENTS | 21 |
| 19.0 | REFER | ENCES | 22 |
| 20.0 | INVES | TIGATOR SIGNATURE | 23 |

# 1.0 ABREVIATIONS AND TERMS

| AE | Adverse Event |
|---|---|
| CFR | Code of Federal Regulations |
| Ch. | Charriere Size of Catheter (also known as French Size) |
| CRF | Case Report Form |
| CRO | Clinical Research Organization |
| GCP | Good Clinical Practice |
| eCRF | Electronic Case Report Form |
| EDC | Electronic Data Capture |
| ePRO | Electronic Patient Reported Outcomes |
| IC | Intermittent Catheter |
| ICH | International Council for Harmonisation |
| ICF | Informed Consent Form |
| IFU | Instructions For Use |
| IRB | Institutional Review Board |
| PHI | Protected Health Information; any information about health status, provision of health care, or payment for health care that can be linked to a specific individual. |
| PI | Principle Investigator |
| SAE | Serious Adverse Event |
| Sponsor | An individual, institution, company, or organization that takes the responsibility to initiate, and manage a clinical trial. For the purposes of this study, the Sponsor is Hollister Incorporated. |
| Study Product | The product being evaluated in the clinical study. For the purposes of this protocol, the Study Product is a single-use hydrophilic intermittent catheter |
| Sub-I | Sub Investigator |
| TMF | Trial Master File |
| UAE | Unexpected Adverse Event |
| USA | United States of America |

#### 2.0 ETHICS

#### 2.1 IRB Review

This non-significant risk clinical study, including the Informed Consent, will be reviewed by an Institutional Review Board (IRB) in accordance with Title 21 of the Code of Federal Regulations (CFR), Parts 50 and 56. Approval by the Board will be obtained prior to the initiation of the study.

This study is considered of minimal risk in that the anticipated risks of harm are no greater, considering probability and magnitude, than those ordinarily encountered in the daily routine of the subjects. This definition is consistent with 21CFR §§ 56.102(i).

#### 2.2 Name and Address of IRB

The study and any amendments will be reviewed by the following IRB:

BRANY IRB (Formerly Asentral IRB)
Biomedical Research Alliance of New York LLC
1981 Marcus Avenue, Suite 210
Lake Success, NY 11042

The IRB above meets the FDA's definition of an Independent Ethics Committee as defined in 21 CFR 812.3(t). Records to support the above statement can be found in the sponsor's Trial Master File (TMF). If additional, or local, IRB approval is required per individual site requirements, records will be stored in the sponsor's TMF.

#### 2.3 Adherence to Ethical Principles

The study will be conducted in accordance with the ethical principles that have their origins in the Declaration of Helsinki.

#### 3.0 INVESTIGATORS AND STUDY ADMINISTRATIVE STRUCTURE

Hollister Incorporated is the Sponsor and financer of this clinical study. The Principal Investigator (PI), Sub-Investigator(s) (Sub-I), and study administrative team (data manager, statistician, etc.) are employees of the Sponsor. Hollister Incorporated is the acting clinical site for this at-home panel study.

#### 3.1 Investigator Responsibilities

It is the responsibility of the PI and Sub-I to follow applicable Good Clinical Practice (GCP) guidelines and regulations including: complying with the protocol procedures, overseeing enrollment of appropriate subjects, addressing subjects' questions or concerns, evaluating and reporting Adverse Events (AE), ensuring Informed Consent is properly obtained, and retaining all study related documents for (or according to local authorities guidelines on record retention) once the study is officially closed.

#### 3.2 Sponsor Responsibilities

It is the responsibility of the sponsor, Hollister Incorporated, to oversee the overall conduct of the clinical study and verify study procedures are adhered to by the Investigator(s). The Sponsor will also maintain accurate product accountability and maintain shipping records for study product. Hollister Incorporated

may transfer any or all trial-related duties and functions to a CRO or vendor, but the ultimate responsibility for the quality and integrity of the study data resides with the sponsor, per ICH Good Clinical Practice 5.2.1.

| <b>4.0</b> Hollist | BACKGROUND/RATIONALE ster Incorporated has developed hydrophilic | technology |
|---|---|---|
| | | Prior to launching |
| | technology, Hollister plans to collect feedback fro | |
| 5.0 | STUDY OBJECTIVES | |
| 5. | The primary Objective of this study is to assess product. Assessment data will be collected to detect technology to be acceptable | hydrophilic technology used on the study letermine whether end users find the hydrophilic |
| | through daily questionnaires intended to track ac | Product safety will also be monitored diverse events. |
| 5. | 5.2 Secondary Objective The secondary objective is to generate evidence | e to support commercial objectives . |
| 6.0 | STUDY PRODUCTS | |
| 6. | The study product Intermittent Catheter marketed by Hollister Incorporated product has been modified Additionally the catheter study participants may not have seen prior. | is a straight, hydrophilic, The original product, The hydrophilic have design enhancements that the |
| | | The study product is packaged as a box of thirty (30). |

individually wrapped, single-use, hydrophilic intermittent catheters.



The study product shall be used with end users who currently use a IC product or have sampled a IC according to protocol procedures, self-catheterize a minimum of IC according to protocol procedures, self-catheterize a minimum of IC according to protocol procedures, self-catheterize a minimum of IC according to protocol procedures, self-catheterize a minimum of IC according to protocol procedures, and are familiar with how to properly use an IC per the Instructions For Use (IFU). This study is considered of minimal risk in that the anticipated risks of harm are no greater, considering probability and magnitude, than those ordinarily encountered in the daily routine of the subjects. This definition is consistent with 21CFR §§ 56.102(i).

The study product to be used in this study is class II devices are those for which general controls alone are insufficient to assure safety and effectiveness, and additional existing methods are available to provide such assurances. Therefore, Class II devices are also subject to special controls in addition to the general controls of Class I devices. Special controls may include special labeling requirements, mandatory performance standards, and post market surveillance. Devices in Class II are held to a higher level of assurance than Class I devices to insure that they will perform as indicated and will not cause injury or harm to patient or user.

# 6.2 Identity of Product, Packaging and Storage, Procedures for Release

| identity of Product, Packaging an | id Storage, Procedures for Release |
|---|---|
| The study product | will be manufactured and released according to the Sponsor's |
| Authorization for Release of Clinical Pr | oduct |
| | The study product |
| shall be manufactured and supplied un | nder Clinical Manufacture Protocol |
| The study product will be labeled | prior to study initiation using the following labels: |



| D. Following completion of steps | , product can be shipped (dispensed) to the subject. | |
|---|---|---|
| Anytime study product is dispensed to a subject Capture (EDC) System on documentation including shipment tracking number | r, research staff will document it in the Electronic Dat Product shipmen bers will also be retained by the sponsor. | |
| • | | |
| | ts after each use, according to their normal practice and theters will be returned to the Sponsor at the end of the provided to them. Sponso in the EDC System on | e |
| as stated in the product IFU. Any unused study casubjects' participation in the study using the will document the date and number of returned ICSTUDY DESIGN The study will be executed at a | theters will be returned to the Sponsor at the end of the provided to them. Sponso | e<br>or |
| as stated in the product IFU. Any unused study casubjects' participation in the study using the will document the date and number of returned IC STUDY DESIGN The study will be executed at a will not require Subjects will be assigned to one of two pocurrently use IC products. Group 2 will included but do use | theters will be returned to the Sponsor at the end of the provided to them. Sponso | e<br>or<br>d<br>o<br>ts |

7.0

| Subjects in Group 2 will be shipped | IC |
|---|---|
| | Subjects will first sample |
| the currently marketed product for a | , or until they use a maximum of 60 Study Catheter |
| whichever occurs first ("sampling period"). After | er the sampling period, subjects will switch to using Study |
| Catheter Subjects will use the study Catheter | for a consecutive , or until they have used |
| all 30 Study Catheter whichever occurs first | . Subjects will be instructed to use both study catheters |
| according to their usual care practices. After ea | nch day, subjects will complete a daily check-in to confirm |
| the number of ICs they have remaining and if the | nere have been changes in their overall health. After using |
| both study catheters, the subjects in Group 2 | will complete an end-of-study questionnaire about their |
| overall experience. | |

#### 8.0 STUDY SUBJECTS

In order to be eligible for participation in this study, each study participant must meet the following inclusion and exclusion criteria.

#### 8.1 Inclusion Criteria for Group 1

Subject who:

- 1. is male and at least 18 years of age
- 2. can speak, read, and write in English
- 3. has been performing unassisted, self-catheterizations, with a Hydrophilic IC, for at least 1 month
- 4. is self-catheterizing
- 5. currently uses a IC and has been for at least 2 weeks
- 6. is willing to provide permission and the means for study staff to contact
- 7. is willing and able to follow the study protocol procedures including completing questionnaires as demonstrated by signing the Informed Consent

#### 8.2 Inclusion Criteria for Group 2

Subject who:

- 1. is male and at least 18 years of age
- 2. can speak, read, and write in English
- 3. has been performing unassisted, self-catheterizations, for at least 1 month
- 4. is self-catheterizing
- 5. currently uses a Hydrophilic IC in hydrophilic IC include but are not limited to:

| 6. | is willing to provide permission and the means for study staff to contact |
|---|---|
| 7. | is willing and able to follow the study protocol procedures including completing online |
| Subject<br>1.<br>2. | questionnaires as demonstrated by signing the Informed Consent sion Criteria for Group 1 t who: is currently undergoing chemotherapy, radiation or steroid therapy has a symptomatic urinary tract infection (UTI) is currently using a product to perform catheterization Performs catheterization |
| Subject<br>1.<br>2. | is currently undergoing chemotherapy, radiation or steroid therapy |
| All sub<br>their he<br>who re<br>study of<br>8.6 Subject | ct Treatment and Care ject care will be consistent with standard health care practices. Subjects will report any changes in ealth status during the course of the study Export health problems may be directed by the PI or designee to seek care from their The PI or designee will follow up with subjects about any that occur until it has resolved for up to after completion. ct Compensation ts will be offered for their participation study. Compensation will be paid out by the Sponsor |
| | subject completing the study procedures. |

## 9.0 STUDY PROCEDURES

| 9.1 | Subject Identification and Recruitment Subjects will be recruited from include but are not limited to: | Possible methods to identify and recruit end users may |
|---|---|---|
| | Once identified as a possible subject, subject will the Sponsor. | be assigned a Study ID by |
| 9.2 | subject will have the opportunity to ask question informed they may end their participation at a | a link to the IRB-Approved, nature and purpose of this study to the subjects. Each ons before deciding whether to participate, and will be ny time. If the subject decides to participate, they will ect is ultimately eligible for the study, the Sponsor will e study product that is mailed to them. |
| 9.3 | Once informed consent is verified, the potenti | al subject will be usion/exclusion eligibility criteria. If a subject meets |
| | enrolled into the study. If the subject does not me be documented within the EDC and the subject w | the subject will be formally neet the screening criteria, the reason for screen-fail will not be enrolled into the study. |

#### 9.4 Method of Assigning Subjects to Study Groups

All subjects will be assigned to one of two possible study Groups. Group 1 will include subjects who currently use IC products. Group 2 will include subjects who currently do not use IC products but do use a different type of IC on the market, as defined in the eligibility criteria in Sections 8.1 and 8.2. Subjects will be assigned either to Group 1 or Group 2 depending on their current IC product reported at time of completing the eligibility screener.

#### 9.5 Blinding

There is no blinding in this study. All study product is open label.

#### 9.6 Prior and Concomitant Therapy

See Sections 8.1 - 8.2 Inclusion Criteria and Sections 8.3 - 8.4 Exclusion Criteria for pertinent prior and concomitant therapy requirements.

#### 9.7 Study Visits and Evaluation Methods

Subjects in Group 1 are enrolled into the study for up to they use their first study product. Subjects are expected to use their typical routine. Study events include completion of electronic ICF, eligibility screening form, baseline form, daily questionnaires, and one end-of-study questionnaire. There are no in-person study visits during this study. Subjects will use and evaluate the study product at their respective homes. Study events for the subjects in Group 1 are summarized below:





completion of electronic ICF, eligibility screening form, baseline form, daily questionnaires, and one endof-study questionnaire. There are no in-person study visits during this study. Subjects will use and evaluate the study product at their respective homes. Study events for the subjects in Group 2 are

summarized below:





#### 9.8 Subject Instructions

| Subjects will be provided | Instructions for Use | |
|---|---|---|
| | | depending on which |
| Group they have been assigned to. The | IFU provided to the subject are based on t | he currently approved |
| IFU for the currently marketed | product. The steps to use Study Cathet | er remain the |
| same as the currently marketed produc | t. The participant study instructions includ | e steps for completing |
| the study procedures/questionnaires a | nd contact information for research staff i | f they experience any |
| issues while participating in the study. | | |

#### 9.9 Compliance

Subjects are expected to fully comply with the protocol procedures and study instructions. If a subject deviates from the protocol at any point, study staff will use to document the event in the EDC system.

The site will be monitored for compliance. If site is found to have multiple deviations, corrective action or re-training may be necessary.

#### 9.10 Subject Withdrawal

Subjects may elect to withdraw from the study at any time for any reason. Data collected up to the point of withdrawal will be eligible for analysis, unless the subject documents in writing to the PI that they refuse use of any and all of their data for analysis. Any new information gained during the study that might affect the subject's desire to continue participation will be conveyed to them in a timely manner. These

procedures are expressed in the ICF that the subject signs. Subjects electing to withdraw from the study are required to return all unused study product.

The Investigator may discontinue a subject from the study at any time without prejudice. Discontinuations are documented on Furthermore, the Sponsor may end the study at any time.

#### **10.0 ADVERSE EVENTS**

An Adverse Event (AE) is any untoward medical occurrence experienced by a subject, which does not necessarily have to be related to the device under investigation. An AE can therefore be any unfavorable and unintended sign, symptom, or disease experienced while also using the device, whether or not considered related to the device.

Based on literature evaluation, expected adverse events that could occur in subjects recruited for this study include:

 These are possible risks with any intermittent catheter usage on the market and are not unique for the study product.

A Serious Adverse Event (SAE) is one that results in death, results in life-threatening illness or injury, requires inpatient hospitalization or prolongation of hospitalization, results in medical intervention to prevent permanent impairment, or results in permanent impairment of body structure or function, or that result in injury or death to a fetus.

• There are no SAE related to the study product anticipated in this study.

An Unanticipated Adverse Event (UAE) occurs when the nature, severity, or frequency of the event is not consistent with the known or foreseeable risk of the anticipated adverse events associated with the study product or procedures involved with this research.

#### 10.1 Handling Adverse Events

Upon study enrollment, all subjects are informed to notify the Investigator immediately if they experience any health or study-related problems. Subjects will be asked daily to report any change in their health status during the course of the study on the Daily Questionnaires

PI or designee will contact the subject if clarification of the information reported on the daily form is needed. The PI will determine if an AE has occurred, the severity of the AE, and if it was related to the study product. AEs will be documented on in the EDC system. Subjects who report AEs may be directed to seek care from their healthcare provider or emergency room, as appropriate.

All AEs are followed to determine resolution for up to by the Investigator and the Adverse Event Form is updated to indicate date of resolution. If at any point, the Investigator determines the subject should no longer remain on the study product, the subject should be discontinued from the study.

#### 10.2 Reporting Adverse Events

Unanticipated Adverse Events (UAE) and Serious Adverse Events (SAE) related to the study product must be reported by the Investigator or Sub-Investigator through the EDC system within documenting on

Investigators are also required to submit a report of SAE to IRB as soon as possible, but in no event later than after the investigator first learns of the event (Guidance for Clinical Practice Adverse Event Reporting to IRBs Improving Human Subject Protection , 2009).

#### 10.3 Study Stopping Rules



#### 11.0 DATA MANAGEMENT

It is the responsibility of the Investigator to ensure the completeness and accuracy of all study data collected in the EDC system. Subject name and contact information will be treated as Protected Health Information and not included in any dataset for analysis. All datasets for study analysis will include only de-identified data.

The electronic ICF and electronic case report forms (eCRFS) will be collected directly from research subjects using a secure, cloud-based EDC and electronic patient reported outcomes (ePRO) system will be configured by the Sponsor Data Manager for study-specific data capture. Study forms such as the Adverse Event Form, Protocol Deviation Form, and Contact Log will be entered by the study personnel at the site.

Subjects will be provided with a link to the EDC/ePRO system via an email, as each study form is made available to them to complete. Subjects will set up their own, secure password to the system and that password remains unknown to the Sponsor. The EDC will provide an audit log that verifies that all ePRO data were entered by the subjects themselves. The audit log will also document when and by whom any modifications were made to the data after initial entry.

To the best of the Sponsor's ability, data logic and validation checks will be configured in the ePRO system so that subjects will receive warning messages at time of entry regarding inconsistent or invalid entries, in order to assure quality and completeness of data. Because the study collects self-report data directly from the study participants, there will be minimal corrections or modifications by the Sponsor to ePRO data. Any modification of any ePRO data will only be done following direct contact and clarification from the research subject. There will be no modification to any data capturing subject opinion or assessment of study product. The Sponsor may contact the subject to clarify factual data, such as date of first study product use, or any unclear responses on the ICF and the Eligibility Screener, to assure proper and full consent of subjects, as well as confirmation of eligibility before study

enrollment. The Sponsor will contact any subject who directly reports or implies a change in their health status, in order to assure subject safety while using the study product.

Access and permissions to the EDC system for data entry, approval signatures, and/or data export are controlled by user identification and password, which are provisioned by the Sponsor. Investigators and other study personnel are trained by the Sponsor in the use of the EDC and application of electronic signatures before the start of the study. The Study Investigator will electronically sign all study data captured in the EDC, prior to data export and analysis.

#### 12.0 STATISTICAL METHODS

#### 12.1 Analysis Principles

Enrolled subjects who provide product assessment data will be eligible for analysis; subjects who screen fail or did not provide any study product assessment data will be excluded from analysis.

#### 12.2 Incomplete Follow-up and Missing Data

In the event that a subject does not complete the full study period, the complete set of data available for that subject prior to loss-to-follow-up will be used for analysis. No imputation of missing data will be performed.

#### 12.3 Multi-Center and Multiple Comparison/Multiplicity Adjustments

Data collected from all study sites will be combined and analyzed as a whole. No multi-center adjustments will be made.

#### 12.4 Sample Size and Power

A sample size of end-users was chosen to attain a margin of error of approximately defect the dropout rate, up to end users will be enrolled to reach a target final sample size of up to

#### 13.0 STATISTICAL ANALYSES

#### 13.1 Primary and Secondary Objective

Study data collected will be analyzed using appropriate statistical methods as defined by the variable's data level (i.e. continuous, ordinal, categorical, etc.). This includes but is not limited to frequency and percentages for categorical measures and mean [standard deviations] for continuous measures.

#### 13.2 Interim Analyses

An interim analysis is planned for when one of the following milestones occur, whichever occurs first: 1) subjects have provided product assessment data via the end of study questionnaire or 2) the study reaches . All subject data that has been gathered and released on or prior to this milestone will be included in the interim analysis.

Any amendments will be documented per Section

#### 14.0 STUDY DOCUMENTATION AND RECORD KEEPING

The Sponsor and clinical site are required to retain essential study documents within a study TMF. The Sponsor is responsible to retain study documentation per the retention schedule set forth in Clinical sites other than Hollister Incorporated are required to retain study documentation for following Sponsor notification of study closure.

#### 15.0 FINAL REPORT

The Sponsor will write and issue an interim report per the schedule provided in Section 13.2 and a final report at study completion. It is the responsibility of the Investigator to provide the interim and final reports to the IRB, as required. In the event that the target sample size is enrolled and available for analysis by the time of the planned interim analysis, a final report will be issued in lieu of an interim report and a note to file will be created to document this event.

#### 16.0 MONITORING

A qualified Hollister Incorporated monitor or designee will monitor the study data to verify that forms are completed, and that the conduct of the trial is in compliance with the currently approved protocol/ amendment(s) procedures, GCP, and any applicable regulatory requirements.

All data collected for this study is subject self-report data via ePRO questionnaire, and therefore there will be no source documents for monitoring. To the best of the Sponsor's ability, data logic and validation checks will be configured in the EDC ePRO module so that subjects will receive warning messages at time of entry about inconsistent or invalid entries, in order to assure quality and completeness of data. Since the study collects there will be minimal corrections or modifications by the Sponsor to ePRO data. Any modification of ePRO data will only be done following direct contact and clarification from the subject. There will be no modification to any data capturing subject opinion or assessment of study product. The Sponsor may contact subjects to clarify factual data, such as date of first study product application, or any unclear responses on the ICF and the Eligibility Screener, to assure proper and full consent of subjects, as well as confirmation of eligibility before study enrollment. The Sponsor will contact any subject who directly reports or implies a change in their health status, in order to assure subject safety while using the study product.

#### 17.0 AMENDMENT PROCEDURES

The Sponsor is responsible for initiating any protocol amendments. The amendments will be reviewed by the PI and approved by the IRB before they are implemented. Investigator(s) are notified of changes, and a copy of the amendment is kept in the TMF.

# **18.0 PROTOCOL ATTACHMENTS**



#### **19.0 REFERENCES**

- 1. FDA. Information Sheet Guidance For IRBs, Clinical Investigators, and Sponsors Significant Risk and Nonsignificant Risk Medical Device Studies https://www.fda.gov/media/75459/download
- 2. FDA. Guidance for Clinical Practice Adverse Event Reporting to IRBs Improving Human Subject Protection . (2009, January). Retrieved from https://www.fda.gov/downloads/regulatoryinformation/guidances/ucm126572.pdf



- ICH Harmonised Guideline for Good Clinical Practice Section 5.2.1. (2015, June 11). Retrieved from
   https://www.ich.org/fileadmin/Public\_Web\_Site/ICH\_Products/Guidelines/Efficacy/E6/E6\_R2\_\_Addendum\_Step2.pdf
- 7. Title 21 of the Code of Federal Regulations Parts 11, 50 54, 56, 812
- 8. World Medical Association. (2018). *Declaration of Helsinki Ethical Principles for Medical Research Involving Human Subjects.*

#### **20.0 INVESTIGATOR SIGNATURE**

I have read the foregoing protocol and agree to conduct the study as outlined herein. Electronic signatures may be used (where possible) in lieu of traditional signatures.